CLINICAL TRIAL: NCT05059158
Title: Amyloid-β Clearance Mechanisms: A Multi-modal Study on Lymphatic, Glymphatic and Blood-brain-barrier Function in Alzheimer's Disease
Brief Title: Amyloid-β Clearance Mechanisms in Alzheimer's Disease
Acronym: AmyClearAD
Status: Recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Robert Perneczky, Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: 18-606; 18-606 (Other Grant/Funding Number: Stiftung Verum); 1081 (Other Grant/Funding Number: Förderung, Forschung und Lehre der LMU;)
Record Dates: First submitted 2021-07-15; First posted 2021-09-28 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer's Disease (AD)
Keywords: Alzheimer's Disease; Mild Cognitive Impairment; Sleep; Actigraphy; Blood-brain-barrier; Amyloid-β Clearance Mechanisms
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Alzheimer's Disease: Patients with a Alzheimer's Disease diagnosis
  Interventions: Radiation: positron emission tomography (PET)
- Mild Cognitive Impairment: Patients with a mild cognitive impairment diagnosis
  Interventions: Radiation: positron emission tomography (PET)
- Subjective Cognitive Decline: Patients with a subjective cognitive decline diagnosis
  Interventions: Radiation: positron emission tomography (PET)

INTERVENTIONS:
Radiation: positron emission tomography (PET) — 18-Flutemetamol PET (clinical indicated) is going to be performed at the visit.

SUMMARY:
The focus of this study is to examine the protein-plaque clearance (Aß) in relation to the blood-brain-barrier, the glymphatic system, brain lymphatic system and enzymatic degradation. In order to achieve this aim the investigators intend to study participants with a Subjective Cognitive Decline, Mild Cognitive Impairment and a mild Alzheimer's disease.

DETAILED DESCRIPTION:
In this study, the investigators want to examine the different mechanisms of the accumulation and the clearance of Aß- deposits with imaging methods. One focus of the study is an improved characterisation of a blood-brain-barrier disorder (which seems to have an impact on the Aß-accumulation). Another main aim is to provide an improved mechanistic clearance model, which integrates crucial components such as the recently proposed cerebral glymphatic and lymphatic pathways, and which addresses the interaction between the different components and their individual contribution to Aβ removal from the brain. A possible connection between sleep and an altered transport mechanism will be analysed. The prospective study cohort (N ~60) will include patients with Mild Cognitive Impairment, mild clinical AD and Subjective Cognitive Decline. All study participants will undergo a detailed clinical and neuropsychological assessment according to a standardised protocol (i.a. MRI, PET, CSF, actigraphy). Follow-up assessments will not be performed in the present project, but are planned in a subsequent study, pending further funding.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of amnestic MCI or AD dementia or clinical normal
* Able to provide written informed consent
* Unchanged pharmacotherapy within 4 days prior to the study specific assessments
* Fluent in German

Exclusion Criteria:

* Unable to give informed consent or has a legal guardian
* Other severe mental disorder, e.g. schizophrenia or bipolar affective disorder
* Clinically relevant depression
* Acute suicidality
* Current alcohol, drug or medication abuse
* History of severe traumatic brain injury within 3 months prior to inclusion
* Structural lesions of the basal ganglia or brain stem
* Severe neurological disorder including (but not limited to) epilepsy, systemic disorders, stroke, repeated transient ischaemic attacks, increased brain intracranial pressure, normal pressure hydrocephalus
* Severe medical disorders including (but not limited to) heart failure, respiratory failure, uncontrolled severe arterial hypertension
* Electronic implants (e.g. cardiac pacemaker) or other MRI contraindication
* Renal failure > stage 3 (GFR < 30 mL/min)
* Pregnancy
* Unresolved malignancies within two years prior to inclusion
* Severe current infections or other chronic or systemic disorders
* Other circumstances which preclude participation based on the investigator's judgement

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SCD, MCI or AD
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Differences in the disruption of the brain-blood-barrier between the subgroups | Baseline
  Name of Measurement: Ktrans; Measurement Tool: DCI sequence (MRI); Unit: min -1
Clearance mechanisms and glymphatic or cerebral lymphatic system | Baseline
  Can a disruption in the cerebral clearance through the glymphatic or cerebral lymphatic system be proven in patients with AD, MCI or SCD?
  Name of Measurement: DTI ALPS; Measurement Tool: DTI MRI; Unit: mean (Dxpro, Dypro)/ mean (Dypro, Dzasc)
Connection between the structural/functional connectivity of the resting networks and the clearance mechanisms | Baseline
  Correlations between correlations of bold fluctuations/ number of tracts and DTI ALPS Index
Differences between sleep and activity in SCD, MCI and AD; Do they have a mediator role in association of the BBB disruption and Aß pathology? | Baseline
  Name of Measurement: Sleep Efficiency, Sleep Time, PIM, TAT, ZCM ;Measurement Tool: Actigraphy; Units: minutes, count
Connection between clinical symptoms, Aß pathology and BBB disorder | Baseline
  Correlations between Clinical Dementia Rating Sum of Boxes, CSF markers (pg/ml) and Aß PET, SUVr and Ktrans map

CONTACTS AND LOCATIONS:
Overall Officials: Robert Perneczky, Prof.Dr.med., Principal Investigator — Klinik und Poliklinik für Psychiatrie und Psychotherapie des LMU Klinikums
Locations (1):
- Klinik und Poliklinik für Psychiatrie und Psychotherapie des LMU Klinikums, München, Bavaria, Germany